CLINICAL TRIAL: NCT03382951
Title: Development and Validation of an Automated Measurement of Child Screen Media Use: FLASH
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); William Marsh Rice University (Other); Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Teresia O'Connor, Associate Professor of Pediatrics, Baylor College of Medicine
Other Study IDs: H-40556; R01DK113269 (NIH)
Record Dates: First submitted 2017-11-29; First posted 2017-12-26 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Sedentary Lifestyle
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy children: Each study is an observational study with no group assignments and no control/placebo.

SUMMARY:
Children's screen media use has been identified as a prominent cause for sedentary time that has been linked to obesity and metabolic syndrome, as well as other unwanted physiologic, psychosocial, and academic outcomes in children. However, no system that is automatic, accurate and unobtrusive has been developed to assess children's screen use on different platforms. Advances in technology, such as person detection, accurate facial recognition based on images, and imaging, computer vision and signal processing algorithms now offer novel and promising solutions to objectively and automatically measure people's screen viewing behaviors. Investigators will leverage these recent advances and integrate them to develop a first of its kind, in-home, unobtrusive, automatic, privacy preserving screen use monitoring system: Family Level Assessment of Screen use in the Home (FLASH) that uses an embedded computing platform connected to a video camera on larger, stationary screens (FLASH-TV); or functions as a background app using a front facing camera (FLASH-Mobile). The trans-disciplinary group, consisting of behavioral researchers at Baylor College of Medicine (BCM) and electrical engineers at Rice University, will develop and asses the validity of the FLASH to accurately identify whether and for how long a child is using screen media devices. In this multiple-PI study, the development of FLASH is led by engineers at Rice. Once a final system has been developed, alpha and beta tested, a validation study will take place in observation labs by the BCM behavioral researchers with 6-11 year old children for FLASH-TV and FLASH-Mobile (n=43). Comparisons of FLASH output will be made to staff observations of children participating in a set of structured predefined activities. Next FLASH will be assessed for feasibility and accuracy for identifying children's screen use across platforms in a naturalistic home setting (n=46), compared to direct observation and screen use diaries. FLASH has the potential of having a significant impact on public health and clinical research regarding screen media use by improving scientist's ability to assess the children's screen use. This can lead to better methodology to understand the impact of screen use on children's health outcomes or intervention effects of screen media reduction programs.

DETAILED DESCRIPTION:
Screen media use and TV viewing has been linked to child obesity through epidemiologic and randomized controlled intervention studies, resulting in excess TV viewing becoming a public health concern. Higher amounts of TV viewing among children have also been associated with decreased fitness and higher risk of metabolic syndrome. While TV viewing has often been used as a marker of sedentary behavior, it has been distinguished from inactivity (or lack of physical activity (PA)), by a meta-analyses that found only a small negative (-0.13) effect size between children's TV viewing and PA. A major limitation of the meta-analyses was most included studies relied on parent or self-report of screen viewing behaviors, potentially introducing errors and under or overestimating the true effect size. Screen media use and TV viewing is a common sedentary behavior among children, and accurate assessment of screen use is important to characterize the role it plays in children's overall sedentary behaviors. Accurate assessment of screen media use and TV viewing is also needed to delineate the causal pathways that screen use plays in children's physical activity, development of obesity, and other health outcomes.

Substantial problems and limitations have been identified in the current available measures of TV viewing, which reduces the likelihood of "high quality exposure assessment" of screen use. The most commonly used measure, child self-report or parent-report to estimate the minutes of TV viewing in a typical day has low correlation (0.27) with home video-observations. The current gold standard method to measure children's TV viewing, direct or video recorded observation, is too expensive and intrusive for most field studies. In addition, it may cause privacy concerns for participants and requires additional costs of coding the video recordings at a later time. TV diaries had higher correlations with home video recording (r=0.84) than parent estimates, but are very burdensome requiring documentation of child activity every 15 min for several days, which may introduce systematic errors. Lastly, children's TV viewing behaviors are quickly changing and many children now view TV shows and movies on other screen devices, such as smartphones and mobile tablets (e.g. iPads or Kindles). In summary, the current ability to measure and monitor how much TV a child watches is intrusive (observations), burdensome (TV diaries) or crude and fraught with error and bias (general estimates). This limits researcher's ability to identify causal associations with health outcomes. While automatic and objective measures of PA, such as accelerometers, have shown validity and reliability for quantifying children's PA, no system that is automatic, accurate and unobtrusive has been developed to assess children's screen use on traditional TV screens or tablets.

Imaging, computer vision and signal processing algorithms have made tremendous progress in the last decade, resulting in high-performance, reliable algorithms for many tasks such as face detection, face recognition, gaze tracking, human activity recognition, and 3D sensing. In collaboration with electrical engineers at Rice University, investigators at Baylor College of Medicine are leveraging these recent advances to build a first-of-its-kind 'Family Level Assessment of Screen use in the Home" (FLASH), a fully integrated, unobtrusive system for accurate, privacy preserving and reliable monitoring of TV and other screen usage by children and adults in their homes. In this study, investigators will focus on (a) Integrating the vision and signal processing algorithms and the imaging hardware required to develop FLASH (Rice investigators); (b) Refining the FLASH hardware and the software pipeline for TVs and mobile devices via alpha and beta laboratory studies (Rice and BCM investigators); (c) Validating the FLASH TV and mobile device against the gold standard (observations) among 6-11 year old children who are old enough to follow instructions in a controlled observation laboratory to ensure fidelity to the protocol (BCM investigators), and (d) Performing a preliminary investigation of the challenges for in-home use and adoption (home feasibility study) (BCM investigators).

The ultimate goal of this project is to develop a highly accurate system to measure the screen use by the index child, across diverse screens, including TVs, smartphones and tablets. Since smartphones and tablets are similar in software and hardware, investigators only need to develop two systems: FLASH-TV and FLASH-Mobile. Both systems will take a three step approach: 1) use detection, 2) index user identification, and 3) usage logging, to assess an index child's screen use. The goal is to merge a child's use across screen platforms into one database to be able to track their screen use across devices along with simultaneous use of devices.

FLASH will be developed collaboratively with electrical engineers at Rice University and behavioral researchers at Baylor College of Medicine in a series of four studies:

STUDY 1: Iterative alpha-tests with small samples of family diads or triads (n=3-5 families per trial) of the individual FLASH components and integrated FLASH systems in the CNRC Metabolic Research Unit (MRU) Observational Lab. Investigators plan for these alpha-tests to occur approximately every 3 months to assess the most recent advances of the FLASH technology. Approximately 3-4 separate alpha test with 3-5 triads per test, resulting in an anticipated sample of 42-60 participants (12-20 triads). The experiences from pilot studies we have conducted, identified that iterative testing of new components with a small sample, followed by refinement and retesting, allows for the ideal tight-loop feedback with input from both teams to capitalize on human subject data collection and allow advancement of the technology development.

STUDY 2: One to six beta tests (depending on results) of the integrated prototype FLASH system with 10 family dyads or triads per test will be conducted also in the CNRC MRU Observational Lab, with a maximum on 240 participants (80 triads or dyads). The experience from the pilot study suggests that data from 10 triads or dyads per beta test will allow adequate assessment of the functionality of the FLASH prototype.

STUDY 3: Lab based validation of the final FLASH-TV and FLASH-Mobile devices in the CNRC MRU Observational Lab with 32 parent-child triads. This number has been revised from our initial estimation based on our experiences in alpha and beta tests. Investigators will recruit 32 parent-sibling triads (96 participants) to complete the validation study. Three of the parent-sibling triads (9 participants) will participate in a pilot study prior to starting data collection on the remaining sample to refine the final validation protocol, if needed. To be conservative, we account for ICC of 0.6 in calculating a sample size required for this validation study. A random sample of 29 subjects who are each measured at least 100 times yields a two-sided 95% confidence interval with a width of 0.25 (margin of error = 0.25/2 = 0.125 = 12.5%) when the estimated ICC is 0.6 as assessed using a two-way mixed-effects ANOVA model.

STUDY 4: Home feasibility study to assess families' willingness to have devices installed in their home for a limited time study period and the ability of the FLASH devices to capture children's screen use across an entire day. With a power of 80% and an alpha of 0.05, to detect a moderate-to large effect (0.4) with bivariate correlation between minutes of TV viewing as measured by FLASH compared to TV diaries a final sample size of 37 families will be needed. A moderate-to-large effect size will help ensure high accuracy for FLASH to measure TV viewing in the home. Investigators anticipate having complete data on 80% of participating families and will therefore recruit 46 families (184 participants, estimating 4 family members per family) to achieve the final sample of 37 families.

Across the four studies, investigators therefore anticipate a total sample size of 448 participants (88 triads in studies 1-3 and 46 families in study 4). Each study is an observational study with no group assignments and no control/placebo.

ELIGIBILITY:
Inclusion Criteria:

* index child 5-11 year old child along with parent (adult 18-65)
* and for some studies a 6-14 years old sibling
* family is fluent in English
* parent willing to allow their children to watch age-appropriate TV or movies and play age-appropriate digital/video games.

Exclusion Criteria:

* Parent or child with a developmental, medical, mental or physical diagnosis (such as Down's syndrome, Autism, psychosis, wheel-chair reliant) that would prevent him/her from following the protocol.

Ages: 5 Years to 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Healthy children living in the greater metropolitan area around the research center
Sampling Method: Non-Probability Sample
Enrollment: 321 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Screen media use/viewing | once, upon enrollment
  Assessment of participant's screen media use as detected by the FLASH system. This will be assessed once per family triad during a task based protocol in the observational labs at the research center compared to staff coding of video/audio recordings of the same time period.

SECONDARY OUTCOMES:
The feasibility to recruit families to test the of the FLASH devices their home | 9 months
  Recruit 30 with at least one 6-11 year old child to use the FLASH on all the screens in their home for at least three days (changes to protocol modifications to barriers posed by pandemic for in-home data collection during several years of study).
The feasibility of the FLASH devices to be used in the family's home | 9 months
  Obtain complete data for three days on 24 families (80%) of the 30 families recruited for the five day study.
The feasibility of the FLASH devices in children's homes to measure the amount of time a child spends viewing TV or other screens | three days
  The FLASH device is capable of capturing the minutes somebody watched a TV, as compared to staff staff labeling of video data in a 60-minute protocol in the child's home.
The feasibility of the FLASH devices in children's homes for future studies | three days
  Participating parents found the FLASH to be acceptable and not excessively intrusive to have in their home

CONTACTS AND LOCATIONS:
Overall Officials: Teresia O'Connor, MD, MPH, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No